CLINICAL TRIAL: NCT03737890
Title: Comparison of Hold Relax Pectoral Stretch & Inspiratory Muscle Training on Pulmonary Function Among Frail Elderly
Brief Title: Hold Relax Pectoral Stretch vs Inspiratory Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U/SERC/92/2018
Record Dates: First submitted 2018-11-07; First posted 2018-11-13 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Function in Frail Elderly

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle Training (Experimental): 4 weeks of inspiratory muscle training
  Interventions: Other: Inspiratory Muscle Training
- Hold Relax Pectoral Stretch (Active Comparator): 4 weeks of hold relax pectoral stretch
  Interventions: Other: Hold Relax Pectoral Stretch

INTERVENTIONS:
Other: Inspiratory Muscle Training — Participants in the experimental group were given Inspiratory Muscle Training by using an IMT device. For this training, the inspiratory load for each participant was set at 30 cmH2O.
  In control group, the participants received 3 sets of passive hold- relax pectoral stretch for each session. Each stretch was maintained for 10 seconds with a rest period of 30 seconds given between the sets.
  Each participant was supposed to complete a total of 12 sessions of exercises, 3 sessions per week for 4 weeks.
  Arms: Inspiratory muscle Training
Other: Hold Relax Pectoral Stretch — In control group, the participants received 3 sets of passive hold- relax pectoral stretch for each session. Each stretch was maintained for 10 seconds with a rest period of 30 seconds given between the sets.
  Each participant was supposed to complete a total of 12 sessions of exercises, 3 sessions per week for 4 weeks.
  Arms: Hold Relax Pectoral Stretch

SUMMARY:
Frailty is a clinical syndrome that alters the structure and function of respiratory system which causes stiffness of thoracic cage and reduces the chest wall compliance in addition of respiratory muscle weakness that can lead to the reduction of pulmonary function. The aim of this study was to compare the effect of inspiratory muscle training (IMT) and hold-relax pectoral stretch on pulmonary function (FVC, FEV1 and FEV1/FVC) among frail elderly

DETAILED DESCRIPTION:
Aging leads to the biological and physiological changes in the human body but it is more pronounced in frail elderly. One of the body systems which will undergo changes due to aging is the respiratory system. Respiratory system changes can be in terms of mechanics, muscular and immunological aspects. These changes often lead to respiratory impairment or more often defined as spirometrically airflow limitation or restrictive- pattern. Aging will change the structure of thoracic cage, causing a reduction in chest wall compliance. Moreover, aging disease such as osteoporosis also causes stiffening of the thoracic cage and kyphosis. As a result, the ribcage is unable to expand and contract, causing difficulty in breathing. In addition, atrophy of skeletal muscles leads to increased loss of lean tissue. With the loss of lean tissue in the respiratory muscles, the pulmonary function of an elderly will subsequently be compromised. All these changes decrease the volume of the thoracic cavity and reduce lung volumes which leads to limitation of air flow, decrease of FEV1, FVC and FEV1/FVC as well as increase in residual volume and functional residual capacity. As a result, elderly will tend to have increased work of breathing compared to younger individuals.

Other than that, immunological changes that occur in the elderly increases their risk of getting respiratory tract infection, leading to development of pulmonary disease such as pneumonia. In addition, elderly have higher exposure to second-hand smoke, toxin exposure from the environment which can predispose them to chronic obstructive pulmonary disease leading to dyspnea and alter the pulmonary function. All these changes can have a strong impact on morbidity, mortality and quality of life in elderly.

As a person ages, observable changes can be seen in body composition and body phenotype. These changes will alter the structure and function of the respiratory system. Prevention and intervention programs are necessary to minimize the loss of respiratory function in order to reverse the progression of frailty condition. Exercises such as inspiratory muscle training (IMT) and hold relax pectoral stretch has been found to be helpful in strengthening the breathing muscles and improving pulmonary function respectively. Studies have shown that these two exercises will help in increasing the pulmonary function but till date there is no study which has been carried out to find the effectiveness of these 2 exercises on pulmonary function in frail elderly.

A total of 34 residents from Seavoy Nursing Home were recruited after screening (excluded; bed ridden participants, not able to communicate and give their consent, suffering from a ruptured eardrum or any other condition of the ear, abnormally low perception of dyspnea, presence of cardiac pacemaker, unable to do overhead movement and hyper-mobility of shoulder). Based on the inclusion criteria, the participants needed to be above 60 years of age, currently residing in a care facility, a citizen of Malaysia, ability to understand Malay, English, Mandarin and Cantonese and able to score more than 16 out of 30 in Montreal Cognitive assessment (MoCA). Score of 16 and above on MoCA was to make sure participants were able to follow and understand the instructions given during testing and intervention. This was followed by assessment for frail criteria. At least 3 of the frail criteria; shrinking, weakness, poor endurance, slowness of gait, and low physical activity level needed to be met by participants. Questions such as body weight, height, losing weight, their daily physical activity, their endurance and power status by self reported exhaustion were asked. For shrinking, body weight and height were measured and compared to nursing homes past 1 year record. Participants with unintentional weight loss of 4.5Kgs or more from past 1 year were considered for this study. Weakness criterion was evaluated by checking the grip strength of the dominant hand with cut-off point for different BMI. Besides that, the poor endurance criterion was assessed using two statements of the CES-D scale: "I felt that everything I did was an effort" and "I could not get going" for much or most of the time, when asked. A low physical activity criterion was met if male scored less than 64 and female less than 52 on Physical Activity Scale for the Elderly (PASE). Besides the slow gait speed criterion was met if the participant took more than 10 seconds to walk back and forth over a ten-foot.

After meeting all the inclusion criteria, participants were randomly divided into either into experimental group who did inspiratory muscle training or control group who did hold-relax pectoral stretch. Pulmonary function (FVC, FEV1, FEV1/FVC) were measured by spirometer in sitting upright position. A nose clip was used and participants were instructed to tightly securing the lips around the mouth piece of spirometer. A single trail was run to make sure participants know how to use the spiromter before actual test was conducted.

For screening purpose, Montreal Cognitive assessment (MoCA) was used to evaluate the cognitive status. Physical Activity Scale for the Elderly (PASE) was used to evaluate the physical activity level of the elderly. Center for Epidemiologic Studies Depression Scale (CES- D) was used to evaluate the poor endurance and energy of the elderly. Dynamometer (Jamar hydraulic hand dynamometer) was used to measure the grip strength of the elderly to evaluate the weakness. Furthermore, Portable spirometer (MIR Spirobank II ®) was used to measure the outcome measures (FVC, FEV1, FEV1/FVC). Last but not least, IMT device (Respironics Threshold IMT) was used for inspiratory muscle training.

34 participants were assigned into two groups; control group and experimental group. Each participant was supposed to complete a total of 12 sessions of exercises, 3 sessions per week for 4 weeks. In control group, the participants received 3 sets of passive hold- relax pectoral stretch for each session. Each stretch was maintained for 10 seconds with a rest period of 30 seconds given between the sets. Participants were in sitting position, shoulders held in abducted position with elbows flexed and both hand joined behind the neck. The subjects were asked to contract the agonist muscles and hold for 10 seconds while resistance was applied to the contraction.

On the other hand, participants in the experimental group were given Inspiratory Muscle Training by using an IMT device (Respironics Threshold IMT). Participants were in Fowler's position. Based on the protocol of Inspiratory Muscle Training, a nose clip was used during the training. Participants were advised to inform the researchers and stop the exercise immediately if they felt dizziness or breathlessness. Before the training, participants were taught how to use the device and were instructed to use the correct breathing technique while using the device. For this training, the inspiratory load for each participant was set at 30 cmH2O. During the protocol, researchers observed the participants for their facial expression to ensure that they do not breath forcefully to exhaust themselves. Verbal cue such as don't lift up the chest when doing the breathing exercise, use diaphragm to perform the exercise were given. Participants performed three sets of ten breaths with resting period of one minute between the sets.

The primary outcome measure in this study was pulmonary function. The measures of pulmonary function were: Forced vital capacity (FVC), forced expiratory volume in one second (FEV1), FEV1/FVC. These were assessed by spirometry and expressed in litres. The measures were assessed with the participants in sitting position with the use of nose clip. A clear instruction was given to the participants to expire forcefully out into the disposable mouthpiece and after the machine provide a sound, the participants were asked to inspire forcefully from the disposable mouthpiece. A trail run was performed before running the actual test. The measurement of FVC, FEV1 and FEV1/FVC was evaluated before and after the intervention. Data was recorded in the data collection sheet. However, during this study there were 2 dropouts from experimental group who refused to continue the exercise after first week of intervention. There were also 2 dropouts from the control group as 1 participant was discharged from the nursing home in the second week of the study and another one felt sick in the last week of intervention. Hence, data analysis was performed only for 15 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* Above 60 years of age
* residing in a care facility
* Able to score more than 16 out of 30 in Montreal Cognitive assessment (MoCA). Score of 16 and above on MoCA was to make sure participants are able to follow and understand the instructions given during testing and intervention.
* At least 3 of the frail criteria (shrinking, weakness, poor endurance, slowness of gait, and low physical activity level)

Exclusion Criteria:

* Low cognitive status (MoCA score less than 16)
* Suffering from a ruptured eardrum or any other condition of the ear
* Severe exacerbations , abnormally low perception of dyspnoea
* Presence of cardiac pacemaker
* Refusal to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | At baseline and after 4 weeks of intervention
Change in Forced Expiratory Volume in 1 Second (FEV1) | At baseline and after 4 weeks of intervention
Ratio of FVC/FEV1 | At baseline and after 4 weeks of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sharma G, Goodwin J. Effect of aging on respiratory system physiology and immunology. Clin Interv Aging. 2006;1(3):253-60. doi: 10.2147/ciia.2006.1.3.253. PMID 18046878
- [Result] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Result] Lowery EM, Brubaker AL, Kuhlmann E, Kovacs EJ. The aging lung. Clin Interv Aging. 2013;8:1489-96. doi: 10.2147/CIA.S51152. Epub 2013 Nov 6. PMID 24235821
- [Result] Keller K, Engelhardt M. Strength and muscle mass loss with aging process. Age and strength loss. Muscles Ligaments Tendons J. 2014 Feb 24;3(4):346-50. eCollection 2013 Oct. PMID 24596700
- [Result] Centers for Disease Control and Prevention (CDC). Vital signs: nonsmokers' exposure to secondhand smoke --- United States, 1999-2008. MMWR Morb Mortal Wkly Rep. 2010 Sep 10;59(35):1141-6. PMID 20829748
- [Result] Vaz Fragoso CA, Gill TM. Respiratory impairment and the aging lung: a novel paradigm for assessing pulmonary function. J Gerontol A Biol Sci Med Sci. 2012 Mar;67(3):264-75. doi: 10.1093/gerona/glr198. Epub 2011 Dec 1. PMID 22138206
- [Result] Pegorari MS, Ruas G, Patrizzi LJ. Relationship between frailty and respiratory function in the community-dwelling elderly. Braz J Phys Ther. 2013 Jan-Feb;17(1):9-16. doi: 10.1590/s1413-35552012005000065. English, Portuguese. PMID 23538454